CLINICAL TRIAL: NCT06806293
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study With an Open-Label Extension to Evaluate the Efficacy, Safety, and Tolerability of Atogepant for the Preventive Treatment of Menstrual Migraine
Brief Title: Study of Oral Atogepant to Assess Adverse Events and Change in Disease Activity in Adult Participants With Menstrual Migraine
Acronym: ATO MM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M24-859; 2024-512946-41 (Other: EU CT)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Menstrual Migraine (MM)
Keywords: Menstrual Migraine; Atogepant; QULIPTA; AQUIPTA
MeSH Terms: interventions — atogepant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atogepant (Experimental): Participant will receive atogepant during Double-Blind period and Open-Label period.
  Interventions: Drug: Atogepant
- Placebo for Atogepant (Placebo Comparator): Participant will receive placebo during Double-Blind period and atogepant during the Open-Label period.
  Interventions: Drug: Atogepant; Drug: Placebo for Atogepant

INTERVENTIONS:
Drug: Atogepant — Oral Tablet
  Other Names: Qulipta; Aquipta
Drug: Placebo for Atogepant — Oral Tablet
  Arms: Placebo for Atogepant

SUMMARY:
A migraine attack is a moderate or severe headache that usually occurs on one side of the head and is often throbbing or pulsating. The headache is often accompanied by sensitivity to light, sensitivity to sound, nausea, or other symptoms. Menstrual migraine (MM) attacks are migraine attacks that occur in individuals before or during their menstrual period. The main goals of the study are to evaluate the efficacy (how well the medicine works), safety, and tolerability (the degree to which any adverse symptoms can be handled by the patients during the study) of atogepant, compared to placebo (looks like the study treatment but has no medicine in it), for the prevention of MM.

Atogepant is an investigational drug being developed for the preventive treatment of menstrual migraine. Participants are randomly assigned to one of the 2 treatment groups called Arms to receive atogepant or matching placebo. There is 1 in a 2 chance for the participant to receive placebo. Approximately 430 adult female participants with menstrual migraine will be enrolled in approximately 85 sites across the world.

Participants will receive oral atogepant or matching placebo for 3 menstrual cycles during the double-blind period. During the open-label treatment period, participants will receive atogepant during each menstrual cycle.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The safety and tolerability of the treatment will be checked by medical assessments, blood tests, checking for adverse events and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* History and eDiary confirmation have regular menstrual cycles within the range of 21 to 35 days in length (Note: menstrual cycle length is calculated as onset of menses until the day before the next onset of menses).
* History of migraine (with or without aura) according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3) for >= 12 months prior to Visit 1/Screening.
* Migraine onset before age 50 years.
* By history at Visit 1/Screening, participant meets ICHD-3 criteria for pure menstrual migraine with or without aura, or menstrually-related migraine with or without aura, i.e., in at least 2 out of 3 cycles, experiences migraine attacks starting during the PMP (Day -2 to Day +3 relative to menses onset) in the opinion of the investigator.
* Participant records 3 perimenstrual periods (PMP) in the eDiary during the screening period, and in at least 2 of 3 PMPs the participant experiences and records a migraine attack in the eDiary with at least 1 migraine day.

Exclusion Criteria:

* History of an average of 15 or more headache days per month during the 3 months prior to Visit 1/Screening per the investigator's judgment, or a current diagnosis of chronic migraine as defined by International Classification of Headache Disorders, 3rd Edition (ICHD-3).
* An average of 15 or more headache days per month recorded in the eDiary during the screening period.
* History of migraine with brainstem aura, hemiplegic migraine, or retinal migraine as defined by ICHD-3.
* Current diagnosis of new persistent daily headache, trigeminal autonomic cephalalgia (e.g., cluster headache), or painful cranial neuropathy as defined by ICHD-3.
* Required hospital/emergency room treatment for migraine attacks 3 or more times within 6 months prior to Visit 1/Screening.
* Presence of other confounding pain syndromes, confounding psychiatric conditions, dementia, epilepsy, or significant neurological disorders other than migraine per investigator judgment.
* Has a condition or situation, which the investigator feels will compromise the safety of the participant or the quality of the data and renders the subject an unsuitable candidate for the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Migraine Days Occurring During the Perimenstrual Period (PMP) | Up to approximately 120 days
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.

SECONDARY OUTCOMES:
Change in Number of Migraine Days (With Moderate or Severe Headache) During the PMP | Up to approximately 120 days
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.
Percentage of Participants Achieving >= 50% Reduction in Number of Migraine Days Averaged Across 3 PMPs | Up to approximately 120 days
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.
Change in Number of Acute Medication Use Days During PMP | Up to approximately 120 days
  An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) for the acute treatment of migraine.
Change in Number of Moderate or Severe Headache Days During PMP | Up to approximately 120 days
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication was used after the start of the headache, in which case no minimum duration will be specified.
Percentage of Participants Achieving 100% Reduction From Baseline in Number of Migraine Days Averaged Across 3 PMPs | Up to approximately 120 days
  A migraine day is defined as any calendar day on which a headache occurs which meets criteria listed, as per participant eDiary.
Percentage of Participants With No Disability/Mild Impairment for 100% of PMP Days As Assessed by Functional Disability Scale (FDS) | Up to approximately 120 days
  FDS is a single item used to measure the participant's level of functional disability.
Change in Number of Headache Days During PMP | Up to approximately 120 days
  A headache day is defined as any calendar day on which headache pain lasting 2 hours or longer occurs unless an acute headache medication was used after the start of the headache, in which case no minimum duration will be specified.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (94):
- China (10):
  - Chinese PLA General Hospital /ID# 267141, Beijing, Beijing Municipality
  - Nanfang Hospital - Southern Medical University /ID# 268510, Guangzhou, Guangdong
  - Hebei General Hospital /ID# 267663, Shijiazhuang, Hebei
  - Renmin Hospital of Wuhan University /ID# 267671, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University /ID# 267885, Suzhou, Jiangsu
  - Shaanxi Provincial PeopleS Hospital /ID# 267827, Xi'an, Shaanxi
  - First Affiliated Hospital of Shanxi Medical University /ID# 267680, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital /ID# 268846, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital /ID# 268511, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine /ID# 267994, Hangzhou, Zhejiang
- Czechia (10):
  - A-Shine s.r.o. /ID# 266048, Pilsen, Plzeň Region
  - Všeobecná Fakultní Nemocnice v Praze /ID# 268100, Prague, Praha 17
  - DADO MEDICAL s.r.o. /ID# 267629, Prague, Praha 2
  - MINKSneuro s.r.o /ID# 267651, Brno
  - Neurologie Brno /ID# 266050, Brno
  - NeuroHK s.r.o. /ID# 266051, Hradec Králové
  - Neuro plus s.r.o. /ID# 266052, Olomouc
  - Clintrial s.r.o. /ID# 266047, Prague
  - Pratia Prague s.r.o. /ID# 268252, Prague
  - Fakultni Thomayerova nemocnice /ID# 266049, Prague
- Germany (9):
  - Neuro Centrum Odenwald - Praxis Erbach /ID# 276171, Erbach im Odenwald, Hesse
  - Studienzentrum Nord-West /ID# 267311, Westerstede, Lower Saxony
  - Universitaetsmedizin Greifswald /ID# 267277, Greifswald, Mecklenburg-Vorpommern
  - Neurozentrum Bielefeld /ID# 276170, Bielefeld, North Rhine-Westphalia
  - Klinikum Ibbenbueren /ID# 267393, Ibbenbueren, North Rhine-Westphalia
  - ZNS Siegen /ID# 268247, Siegen, North Rhine-Westphalia
  - Pharmakologisches Studienzentrum Chemnitz GmbH /ID# 267285, Chemnitz, Saxony
  - Ambenet Hausarztpraxis /ID# 267309, Leipzig, Saxony
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 267310, Berlin
- Hungary (8):
  - MIND Clinic /ID# 267652, Budapest
  - Cortex Study Center /ID# 266639, Budapest
  - Clinexpert Kft /ID# 266644, Budapest
  - Semmelweis Egyetem /ID# 266636, Budapest
  - Semmelweis Egyetem /ID# 266752, Budapest
  - UNO Medical Trials /ID# 266643, Budapest
  - S-Medicon Kft /ID# 266637, Budapest
  - Uzsoki Utcai Kórház /ID# 266641, Budapest
- Italy (9):
  - Azienda Ospedaliero Universitaria Careggi /ID# 276163, Florence, Firenze
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 267062, Milan, Milano
  - Istituto Auxologico Italiano - Ospedale San Luca /ID# 276161, Milan, Milano
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli /ID# 267023, Naples, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 266859, Rome, Roma
  - ICOT Istituto Marco Pasquali /ID# 267288, Latina
  - Fondazione Mondino Istituto Neurologico Nazionale a Carattere Scientifico IRCCS /ID# 267922, Pavia
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 267926, Perugia
  - ASU FC - P.O. Universitario Santa Maria della Misericordia /ID# 267019, Udine
- Japan (10):
  - Konan Medical Center /ID# 266867, Kobe, Hyōgo
  - Fujitsu Clinic /ID# 266877, Kawasaki-shi, Kanagawa
  - Umenotsuji Clinic /ID# 266834, Kochi, Kochi
  - Sendai Headache and Neurology Clinic Medical Corporation /ID# 266864, Sendai, Miyagi
  - Ooba Clinic For Neurosurgery & Headache /ID# 266866, Ōita, Oita Prefecture
  - Chibune General Hospital /ID# 266874, Osaka, Osaka
  - Tominaga Clinic - Osaka /ID# 268228, Osaka, Osaka
  - Usuda Clinic Of Internal Medicine /ID# 266870, Setagaya-ku, Tokyo
  - Tokyo Headache Clinic /ID# 266863, Shibuya-ku, Tokyo
  - Nagaseki Headache Clinic /ID# 266865, Kai, Yamanashi
- Poland (8):
  - Solumed Centrum Medyczne /ID# 267220, Poznan, Greater Poland Voivodeship
  - Athleticomed Sp. z o.o /ID# 266434, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - SPZOZ Szpital Uniwersytecki w Krakowie /ID# 266443, Krakow, Lesser Poland Voivodeship
  - Instytut Zdrowia Dr Boczarska Jedynak /ID# 266073, Oświęcim, Lesser Poland Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 266732, Gdansk, Pomeranian Voivodeship
  - Novo-Med Zielinski i wspolnicy SP. J. /ID# 266433, Katowice, Silesian Voivodeship
  - Neuro-Care Sp. z o.o. sp.k /ID# 267883, Katowice, Silesian Voivodeship
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak /ID# 266437, Wroclaw
- Portugal (10):
  - Unidade Local de Saude do Alto Ave, EPE /ID# 266168, Guimarães, Braga District
  - Hospital da Luz /ID# 266182, Lisbon, Lisbon District
  - Unidade Local de Saude de Loures-Odivelas, EPE /ID# 266190, Loures, Lisbon District
  - Unidade Local de Saude de Matosinhos, EPE /ID# 266170, Senhora da Hora, Porto District
  - Unidade Local de Saude de Almada-Seixal, EPE /ID# 276215, Almada, Setúbal District
  - Unidade Local de Saude da Regiao de Aveiro, EPE /ID# 266187, Aveiro
  - 2CA-Braga, Hospital de Braga /ID# 276218, Braga
  - Unidade Local de Saude de Santa Maria, EPE /ID# 275932, Lisbon
  - Unidade Local de Saude Sao Joao, EPE /ID# 266185, Porto
  - Unidade Local de Saude da Arrabida, EPE /ID# 266183, Setúbal
- South Korea (5):
  - Hallym University Dongtan Sacred Heart Hospital /ID# 267473, Hwaseong, Gyeonggido
  - Nowon Eulji Medical Center, Eulji University /ID# 267474, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 267477, Seoul, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital /ID# 267475, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 267476, Seoul, Seoul Teugbyeolsi
- Spain (4):
  - Hospital Clinic de Barcelona /ID# 276468, Barcelona
  - Hospital Clinico San Carlos /ID# 275896, Madrid
  - Hospital Universitario La Paz /ID# 276332, Madrid
  - Hospital Clinico Universitario de Valladolid /ID# 275899, Valladolid
- Taiwan (5):
  - China Medical University Hospital /ID# 266423, Taichung
  - National Cheng Kung University Hospital /ID# 267754, Tainan
  - Mackay Memorial Hospital /ID# 266421, Taipei
  - Taipei Veterans General Hospital /ID# 266418, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 266424, Taoyuan
- United Kingdom (6):
  - Royal Sussex County Hospital /ID# 268362, Brighton, East Sussex
  - St Pancras Clinical Research /ID# 268653, London, Greater London
  - Guy's Hospital /ID# 267587, London, Greater London
  - Breckland Alliance /ID# 268772, Thetford, Norfolk
  - Oxford University Hospitals - John Radcliffe Hospital /ID# 267659, Oxford, Oxfordshire
  - The Adam Practice /ID# 268116, Poole

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-859